CLINICAL TRIAL: NCT04805606
Title: A Randomized, Open-label, and Parallel Study to Assess Pharmacokinetic/Pharmacodynamic Profiles and Safety of CKD-843 in Male Volunteers
Brief Title: A Clinical Traial to Assess Pharmacokinetic/Pharmacodynamic Profiles and Safety of CKD-843
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A107_01PK2012
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Sequence 1 (Experimental): CKD-843 A - 27mg, Single Dose
  Interventions: Drug: CKD-843 A
- Sequence 2 (Experimental): CKD-843 A - 45mg, Single Dose
  Interventions: Drug: CKD-843 A
- Sequence 3 (Experimental): CKD-843 A - 56mg, Single Dose
  Interventions: Drug: CKD-843 A
- Sequence 4 (Experimental): CKD-843 B - 45mg, Single Dose
  Interventions: Drug: CKD-843 B
- Sequence 5 (Active Comparator): CKD-843-R
  Interventions: Drug: CKD-843-R

INTERVENTIONS:
Drug: CKD-843 A — Single Dose
  Arms: Sequence 1; Sequence 2; Sequence 3
Drug: CKD-843 B — Single Dose
  Arms: Sequence 4
Drug: CKD-843-R — QD, PO
  Arms: Sequence 5

SUMMARY:
A Clinical Traial to Assess Pharmacokinetic/Pharmacodynamic Profiles and Safety of CKD-843

DETAILED DESCRIPTION:
A Randomized, Open-label, and Parallel Study to Assess Pharmacokinetic/Pharmacodynamic Profiles and Safety of CKD-843 in Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Those who aged between 19 to 50 inclusion of man who concerned about androgenic alopecia.
* Those who has body weight ≥ 50kg.
* Those who has calculated body mass index(BMI) of 18.5 ≤ ~ < 27.0 kg/m2

  * Body Mass Index, kg/m2= Body weight(kg)/[Height(m)2]
* Those who consent to proper contraception and do not donate sperm until 6 months after the last administration of investigational product.
* Those who understanding the detailed description of this clinical trial and voluntarily decide to participate.

Exclusion Criteria:

* Those who have clinically significant disease or medical history of Hepatopathy, Renal dysfunction, Neurological disorder, Immunity disorder, Respiratory disorder, Genitourinary system disorder, Hemato-oncology disorder, Cardiovascular disorder or Psychical disorder
* Those who have history of hypersensitivity to active pharmaceutical ingredient, 5α-reductase inhibitor, tocopherol.
* Those who have the screening(D-28~D-2) test results written below

  * AST, ALT > 1.25 times higher than upper normal level
  * Total bilirubin > 1.5 times higher than upper normal level
  * eGFR (estimated Glomerular Filtration Rate, which is calculated by MDRD) < 60 mL/min/1.73m2
  * "Positive" or "Reactive" test result of Hepatitis B & C, HIV, RPR
  * Under 5 min resting condition, systolic blood pressure >150 mmHg or <90 mmHg, diastolic blood pressure >100 mmHg or <50 mmHg
* Those who have a drug abuse history within one year or positive reaction on urine drug screening test.
* Those who received following drugs, which may affect results of clinical trial and safety Ethical-the-counter (ETC) drugs and herbal medicines within 14 days before the first administration and Over-the-counter (OTC) drugs, health foods and vitamin preparations within 7 days before the first administration of the investigational product.
* Those who take barbiturate and related (causing induction or inhibition of metabolism) drug within 30 days before the first administration of investigational product.
* Those who exceeding smoke consumption criteria or can't stop smoking during hospitalization period.

  * Criteria: Smoke > 10 cigarettes/day
* Those who exceeding an alcohol and caffeine consumption criteria or can't stop consuming alcohol and caffeine during hospitalization period.

  * Criteria: Caffeine > 5 cups/day, Alcohol > 210 g/week
* Those who took grapefruit within 7 days before the first administration of investigational product.
* Those who received investigational product by participating in other clinical trial within 6 months before the first administration of investigational product.
* Those who donated whole blood within 60 days or apheresis within 30 days before the first administration of investigational product.
* Those who received transfusion within 30 days before the first administration of investigational product.
* Those who are deemed inappropriate to participate in clinical trial by investigators.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
AUClast of CKD-843 A, CKD-843 B | Day 1(Pre-dose(0 hour), 2, 4, 8 12 hours)
  Area under the concentration-time curve from time zero to last
AUCinf of CKD-843 A, CKD-843 B | Day 1(Pre-dose(0 hour), 2, 4, 8 12 hours)
  Area under the concentration-time curve from zero up to ∞
AUC0-90days of CKD-843 A, CKD-843 B | Day 1(Pre-dose(0 hour), 2, 4, 8 12 hours)
  Area under the concentration-time curve from time zero to 90 days
AUClast of CKD-843-R | Day 1(Pre-dose(0 hour), 1, 2, 3, 4, 6, 8, 10, 12 hours)
  Area under the concentration-time curve from time zero to last
AUCinf of CKD-843-R | Day 1(Pre-dose(0 hour), 1, 2, 3, 4, 6, 8, 10, 12 hours)
  Area under the concentration-time curve from zero up to ∞
AUC0-90days of CKD-843-R | Day 1(Pre-dose(0 hour), 1, 2, 3, 4, 6, 8, 10, 12 hours)
  Area under the concentration-time curve from time zero to 90 days

SECONDARY OUTCOMES:
Tmax of CKD-843 A, CKD-843 B | Day 1(Pre-dose(0 hour), 2, 4, 8 12 hours)
  Time to maximum plasma concentration
t1/2 of CKD-843 A, CKD-843 B | Day 1(Pre-dose(0 hour), 2, 4, 8 12 hours)
  Terminal elimination half-life
CL/F of CKD-843 A, CKD-843 B | Day 1(Pre-dose(0 hour), 2, 4, 8 12 hours)
  Apparent clearance
Vd/F of CKD-843 A, CKD-843 B | Day 1(Pre-dose(0 hour), 2, 4, 8 12 hours)
  Apparent volume of distribution
Tmax of CKD-843-R | Day 1(Pre-dose(0 hour), 1, 2, 3, 4, 6, 8, 10, 12 hours)
  Time to maximum plasma concentration
t1/2 of CKD-843-R | Day 1(Pre-dose(0 hour), 1, 2, 3, 4, 6, 8, 10, 12 hours)
  Terminal elimination half-life
CL/F of CKD-843-R | Day 1(Pre-dose(0 hour), 1, 2, 3, 4, 6, 8, 10, 12 hours)
  Apparent clearance
Vd/F of CKD-843-R | Day 1(Pre-dose(0 hour), 1, 2, 3, 4, 6, 8, 10, 12 hours)
  Apparent volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: MinSoo Park, M.D. Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No